CLINICAL TRIAL: NCT02156089
Title: Neuroimaging Omega-3 and Reward in Adults With ADHD (NORAA) Trial
Brief Title: Neuroimaging, Omega-3 and Reward in Adults With ADHD (NORAA) Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: 140120; 14-AA-0120
Record Dates: First submitted 2014-06-04; First posted 2014-06-05 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12-21

CONDITIONS: Attention Deficit Disorder; Attention Deficit Hyerpactivity Disorder
Keywords: fMRI; Reward Processing; Nutrition; Omega-3 Fatty Acids; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Other: Highly unsaturated omega-3 fatty acids — Nitrient - Matched Placebo of 3 g/d of macademia nut oil (in comparison to 3 g/d of omega-3 highly unsaturated fatty acids).

SUMMARY:
Background:

- People with attention-deficit hyperactivity disorder (ADHD) often have problems with motivation and rewards. . Omega-3 fats have helped symptoms of ADHD improve in children. Researchers want to learn more about the brain activity of people with ADHD and see how taking omega-3 fats might help.

Objective:

- To learn more about how omega-3 fats affect brain activity and ADHD symptoms.

Eligibility:

- Adults age 18 55 with ADHD symptoms.

Design:

* Participants will be screened with medical history and review of medical records.
* For study visit 1, participants will have a medical examination and be interviewed to confirm they have ADHD. They will have an IQ test and give blood and urine samples. Height, weight, and blood pressure will be measured. They will also need to sign consent to agree to take part in the study. They will be asked to complete a food diary for 4 days
* For visit 2, participants will give a blood sample. They will complete questionnaires about their mood and ADHD symptoms.. They may give a blood or saliva sample for genetic testing.
* Participants will have a magnetic resonance imaging (MRI) scan. They will lie on a table that slides in and out of a metal cylinder. It makes loud noises; participants will get earplugs. This scan examines the structure of the brain.
* Participants will have a functional MRI scan. This scan measures the function of the brain while the volunteer is performing tasks in the scanner. They will stop ADHD medications 48 hours before this scan.
* Participants will receive key-lime flavored omega-3 smoothie mix or placebo to takeevery day
* For visit 3, participants will give blood samples and complete questionnaires.
* For visit 4, participants will be weighed and have a blood test and MRI scans as per before. They will repeat the questionnaires and will guess whether they received the omega-3 or placebo.

DETAILED DESCRIPTION:
Objective:

Both attention deficit hyperactivity disorder (ADHD) and addictive behaviors have been persistently related to impaired reward-related processes in the ventral striatum as evidenced by functional magnetic resonance imaging studies (fMRI). These impairments characterized by decreased BOLD activation are thought to be linked to dopamine pathways including decreased D2 receptor function. Omega-3 highly unsaturated fatty acids (HUFAs) are critical for cell-signaling among other complex functions throughout the central nervous system. Animal models have demonstrated that depriving animals of the omega-3 DHA in utero significantly decreases the density of ventral striatal D2- like receptors and furthermore depletes dopamine in the nucleus acumens by 40-60%. The behavioral profile of animals subjected to dietary induced deficiencies of omega-3 reflect decreased goal-directed behavior and increased goal-irrelevant activity, hyperactivity, increased anxiety and reduced behavior flexibility. Abnormally low levels of omega-3 HUFAs have been persistently reported in the erythrocytes of both children and adults with ADHD while supplementation with omega-3 HUFAs was found in a meta-analysis of 10 clinical trials to improve symptoms of ADHD. However, to date no one has tested the potential mediating effects of omega-3 supplementation in reward-related processes in adults with ADHD using neuroimaging techniques. There is hence a need to research the potential treatment effects of omega-3 on assessments of brain function. Therefore, the primary objective of this study is to test the effects of omega-3 intervention (compared to a placebo) in increasing ventral striatal activation during the monetary incentive delay (MID) task. Secondary objectives include collecting neuroimaging data and standardized questionnaires measuring, mood, quality of life and symptoms of ADHD.

Study Population:

150 adults, other-wise healthy, aged 18-55 with ADHD.

Design:

The active group will be stratified according to age and sex to either an active intervention group receiving (1) 3000 mg of omega-3 HUFA smoothie or a placebo group (2) 3000 mg of smoothie macadamia nut oil for 16 weeks. After enrollment and baseline testing, active participants will be randomized to either the treatment or placebo group and instructed to begin consumption of assigned emulsions. Randomized participants will be assessed at baseline, 1 month, 8 weeks, and 16 weeks.

Outcome Measures:

The primary outcome assessments will measure ventral-striatum activation during the MID task. Secondary objectives include: structural MRI, symptoms of ADHD using the Conner s Adult ADHD Rating Scales; negative affective symptoms; endocannabinoid levels and weight change.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be 18 or over and up to 55 years old.

* In general good health.
* Body Mass Index (BMI) between 18 and 35.
* Able to come to the NIH clinical center for each of their scheduled appointments for the duration of the study and have a working phone number.
* Able to understand the consent form and provide written informed consent.
* Have an IQ of 70 or greater as assessed by the WASI for fast IQ testing (a score of less than this is considered to have global intellectual disability - classified in DSM-IV as mental retardation). There are often issues around the ability to give informed consent in adults with global intellectual disability.
* Meet DSM diagnostic criteria for ADHD as assessed by the CAADID Conners Adult ADHD Diagnostic Interview for DSM-IV.
* Have significant symptoms of ADHD despite concurrent pharmacological and psychological therapies as assessed by the Connors Adult ADHD rating scale (CAARS) (as assessed at telephone screen).
* Be willing to have a 48hour wash-out of stimulant medication prior to both baseline and follow-up scans.
* Willing to stop all nutritional supplements including omega-3 fats.
* Willing to stop eating seafood for the study duration of 16 weeks.
* Be willing to have 2 MRI scanning sessions.
* People who are willing to take the smoothie emulsion every day for 16 weeks.

EXCLUSION CRITERIA:

* Any medical illness or treatment that in the view of the investigators would compromise participation in research or participant safety, as determined by medical history, physical examination, laboratory tests (see details under Screening measures below), including, but not limited to:
* Unstable medical conditions requiring immediate intervention.
* Unstable or rapidly progressive neurological diseases.
* History hemorrhagic or ischemic stroke within the last 3 months.
* Known heart disease.
* Hypertension.
* Asthma
* If the participant is related to the study investigator or their superior, subordinate, or immediate family member.
* HIV positive.
* Significant dietary limitations:

Allergy, hypersensitivity, or intolerance to fish oils or omega-3 fats which are found in fish..

* Allergy, hypersensitivity, or intolerance to Macadamia nuts or any nuts such as almonds, walnuts, pecans, peanuts, etc.
* Pregnancy or breastfeeding (by urine pregnancy test; self-report).
* Reported consumption of fish and seafood three or more times per week within the last three months.
* Regular consumption of omega-3 supplements (e.g., cod liver oil, borage oil, fish oil or evening primrose oil) , defined as an average of 250 mg/day of omega-3 HUFAs over the previous 3 months.
* Severe alcohol or substance use disorder according to the AUDIT.
* Acute intoxication or withdrawal from alcohol or other CNS active substances to the extent that they may impair capacity to provide informed consent or participate in research.
* Some neuropsychiatric disorders are either so rare or associated with such profound alterations of brains structure and function that they will be excluded. This includes a diagnosis of severe Bipolar disorders or Axis 1 psychotic disorder assessed by SCID, including schizophrenia, psychosis NOS, autism, substance dependence; dementia, eating disorder.
* Cognitive impairment severe enough to preclude informed consent or valid responses on self-report questionnaires.
* Behavioral instability significant enough to impair ability for consent and participation.
* Participation in other research studies that in the opinion of the investigators would interfere with study outcomes or study compliance.
* On any of the following medications: Atomoxetine (Strattera), bupropion (Wellbutrin), tricyclic antidepressants (imipramine), alpha adrenergic agonists (clonidine, guanfacine) or modafinil (Provigil) depending whether dose interferes with scan and whether or not patient can stay on same dose throughout study.
* Use of non-steroidal anti-inflammatory drugs (NSAIDs), dalteparin, dipyrdamole, enoxaparin, ticlopedine, more than once per week within the last three months.
* Living situation unsuitable for the storage or use of intervention materials.

MRI Exclusion Criteria:

* Have ferromagnetic objects in their bodies, which might be adversely affected by MRI (e.g., surgical clips, metal fragments in or near brain, eye or blood vessels, cardiac or neurological pacemaker, cochlear or eye implant). Any doubt about presence of these objects will result in exclusion from this study.
* Extreme claustrophobia.
* Left-handed individuals.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2014-06-04; Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
To test if omega-3 HUFA intervention results in greater ventral-striatal activation during a reward task in adults with ADHD compared to a placebo group between baseline and follow up at 16 weeks. | baseline and afte 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Hibbeln, M.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bondi CO, Taha AY, Tock JL, Totah NK, Cheon Y, Torres GE, Rapoport SI, Moghaddam B. Adolescent behavior and dopamine availability are uniquely sensitive to dietary omega-3 fatty acid deficiency. Biol Psychiatry. 2014 Jan 1;75(1):38-46. doi: 10.1016/j.biopsych.2013.06.007. Epub 2013 Jul 25. PMID 23890734
- [Background] Zimmer L, Delion-Vancassel S, Durand G, Guilloteau D, Bodard S, Besnard JC, Chalon S. Modification of dopamine neurotransmission in the nucleus accumbens of rats deficient in n-3 polyunsaturated fatty acids. J Lipid Res. 2000 Jan;41(1):32-40. PMID 10627499
- [Background] Zimmer L, Delpal S, Guilloteau D, Aioun J, Durand G, Chalon S. Chronic n-3 polyunsaturated fatty acid deficiency alters dopamine vesicle density in the rat frontal cortex. Neurosci Lett. 2000 Apr 21;284(1-2):25-8. doi: 10.1016/s0304-3940(00)00950-2. PMID 10771153